CLINICAL TRIAL: NCT01513226
Title: Cycled Light Exposure Reduces Fussing and Crying in Very Preterm Infants
Brief Title: Cycled Light and Crying of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CH-160.7.002.920-3
Record Dates: First submitted 2012-01-11; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Crying; Sleep
Keywords: cycled light; dim light; circadian rhythm; actigraphy, sleep; premature infant
MeSH Terms: conditions — Crying; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dim light (Experimental): Day and nighttime dim light conditions
  Interventions: Other: Cycled light

INTERVENTIONS:
Other: Cycled light — lights on at daytime, lights off at nighttime

SUMMARY:
This study shows that cycled light during neonatal care reduces infant's fussing and crying behavior at 5 and 11 weeks corrected age and improves growth during neonatal care.

ELIGIBILITY:
Inclusion Criteria:

* very preterm infants (≤ 32 0/7 weeks gestational age, GA)

Exclusion Criteria:

* major cerebral injuries such as intraventricular haemorrhage grade III (according to Papile 16) or periventricular leukomalacia or venous infarction (according to Govaert and de Vries 17) diagnosed by cranial ultrasound
* retinopathy of prematurity grade III and IV
* congenital malformations
* small for gestational age (birth weight < 3rd percentile)
* prenatal infections
* intrauterine drug exposure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
mean duration and change over time for total duration per 24 hours for crying variables | 5 and 11 weeks corrected age
  mean duration per 24 hours for following variables: content, fussing, crying, unsoothable crying change over time, measured at 5 and 11 weeks corrected age
  measured by diary

SECONDARY OUTCOMES:
mean sleep duration per 24 hours and change over time | 5,11 and 25 weeks corrected age
  mean sleep duration per 24 hours measured by sleep diary measured at 5, 11 and 25 weeks corrected age, for adressing change over time
mean weight gain per day | during hospital stay
  mean weight gaing per day during hospital stay.
mean activity count per 24 hours and change over time | 5, 11, and 25 weeks corrected age
  mean activity count per 24 hours measured by actigraph recordings measured at three time points, 5, 11 and 25 weeks corrected age to adress change over time

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Jenni, MD, Principal Investigator — Children's Hospital Zurich

REFERENCES:
- [Derived] Guyer C, Huber R, Fontijn J, Bucher HU, Nicolai H, Werner H, Molinari L, Latal B, Jenni OG. Very preterm infants show earlier emergence of 24-hour sleep-wake rhythms compared to term infants. Early Hum Dev. 2015 Jan;91(1):37-42. doi: 10.1016/j.earlhumdev.2014.11.002. Epub 2014 Nov 27. PMID 25460255
- [Derived] Guyer C, Huber R, Fontijn J, Bucher HU, Nicolai H, Werner H, Molinari L, Latal B, Jenni OG. Cycled light exposure reduces fussing and crying in very preterm infants. Pediatrics. 2012 Jul;130(1):e145-51. doi: 10.1542/peds.2011-2671. Epub 2012 Jun 11. PMID 22689866